CLINICAL TRIAL: NCT02970110
Title: Specimen Collection Study for H. Pylori Testing in Patients With Dyspepsia
Brief Title: Specimen Collection Study for H. Pylori Testing
Status: Completed | Type: Observational
Sponsor: Biomerica (Industry)
Responsible Party: Sponsor
Other Study IDs: HPY-COL-001
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Helicobacter Infections
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to acquire human specimens from subjects undergoing routine endoscopy with gastric biopsy for the diagnosis of active H. pylori infection.

DETAILED DESCRIPTION:
This is a prospective study designed to acquire and bank human specimens from subjects who are scheduled for routine upper endoscopy for symptoms such as dyspepsia. This study will be conducted at a minimum of 2 sites in the United States. Investigator sites will enroll prospective subjects who meet the inclusion / exclusion criteria. A case report form (CRF) provided by the sponsor will be used to capture basic demographic information (DOB, age, gender, race/ethnicity), medication history, and related clinical information. The CRFs will also record the results of the following tests performed with the gastric biopsy tissue specimens: histology and rapid urease test (RUT).

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 and to 75 years.
* Able to read, speak, and understand English or have access to a translator in subject's native language.
* Patients without prior H. pylori eradication treatment.
* Currently not on proton pump inhibitors, antibiotics or bismuth

  * Discontinuation at least 2 weeks prior to endoscopy and specimen collection.
* Present with signs and symptoms of dyspepsia [e.g. upper abdominal discomfort or pain]
* Undergo gastric biopsies as part of routine care
* Physician able to provide histology and rapid urease result on biopsy specimens.

Exclusion Criteria:

* Aged less than 21 years old or older than 75 years
* Unable to provide consent.
* Patients with a history of prior H. pylori eradication therapy.
* Currently on proton pump inhibitors, antibiotics or bismuth and cannot or will not discontinue
* Previous upper gastrointestinal surgery, such as bariatric surgery, Nissen fundoplication, or Roux-en-Y.
* Any unstable or poorly-controlled medical or psychiatric condition.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects scheduled for routine upper endoscopy for upper gastrointestinal tract symptoms such as dyspepsia. All prospective subjects must be off of proton-pump inhibitors, antibiotics, and bismuth for at least 2 weeks prior to submission of the stool specimen and undergoing endoscopy.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Non-invasive collection procedure | 1 year
  This study is designed to collect specimens to supplement repository specimens for product validation purposes. The endoscopy results and specimens will be used in a future clinical trial of a non-invasive in vitro diagnostic assay for the detection of H. pylori antigen. institutional review board approval is sought in order to be able to use human specimens for validation of in vitro diagnostics.

CONTACTS AND LOCATIONS:
Overall Officials: James R Buxbaum, M.D., Principal Investigator — University of Southern California, Los Angeles County Hospital
Locations (4):
- United States (4):
  - Del Sol Research Management, Inc., Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Medley Research Associates, Medley, Florida
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Demographics including age, gender, geographical location, histology and RUT results collected in this study will be shared with researchers involved with a future evaluation of an in vitro diagnostic device product in development at Biomerica.